CLINICAL TRIAL: NCT04626973
Title: Effects of Ezetimibe Combination Therapy for Patients With Atherosclerotic Cardiovascular Disease; Randomized Comparison of LDL-cholesterol Targeting <70 Versus <55mg/dL; Ez-PAVE Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0903
Record Dates: First submitted 2020-10-20; First posted 2020-11-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Dyslipidemia; ASCVD; Coronary artery disease
MeSH Terms: conditions — Atherosclerosis; Dyslipidemias; Coronary Artery Disease | interventions — Ezetimibe; Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Intervention Model Description: At the time of enrollment, we will stratify all patients according to LDL-cholesterol <100mg/dL, DM, and acute coronary syndrome, and randomly assign them in two groups according to LDL-cholesterol targeting level with a 1:1 ratio: "Intensive-targeting group" vs. "Conventional-targeting group". In addition, patients in each group will be randomly assigned to receive two lipid-lowering therapy regimen with a 1:1 ratio: "Ezetimibe/Statin combination therapy" vs. "Statin monotherapy".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive-targeting group (Experimental)
  Interventions: Drug: Ezetimibe/Statin Combination therarpy (ezetimibe plus rosuvastatin); Drug: Statin monotherapy (rosuvastatin or atorvastatin)
- Conventional-targeting group (Active Comparator)
  Interventions: Drug: Ezetimibe/Statin Combination therarpy (ezetimibe plus rosuvastatin); Drug: Statin monotherapy (rosuvastatin or atorvastatin)

INTERVENTIONS:
Drug: Ezetimibe/Statin Combination therarpy (ezetimibe plus rosuvastatin) — For statin naive patients, patients would initially receive Ezetimibe 10mg plus Rosuvastatin 10 or 20 mg.
  For non-statin naive patients, regimens are to be changed to the equivalent dose of ezetimibe+rosuvastatin combination in case of already achieved LDL-cholesterol target (<55 mg/dL) and to be dosed up than the equivalent dose of study drugs in case of not yet achieved LDL-cholesterol target.
  Arms: Intensive-targeting group
Drug: Statin monotherapy (rosuvastatin or atorvastatin) — For statin naive patients, patients would initially receive Rosuvastatin 20mg or Atorvastatin 40 or 80 mg.
  For non-statin native patients, regimens are to be change to equivalent dose of atorvastatin or rosuvastatin in case of already achieved LDL-cholesterol target (<55 mg/dL) and to be dosed up than the equivalent dose of study drugs in case of not yet achieved LDL-cholesterol target.
  Arms: Intensive-targeting group
Drug: Ezetimibe/Statin Combination therarpy (ezetimibe plus rosuvastatin) — For statin naive patients, patients would initially receive Ezetimibe 10mg plus Rosuvastatin 5 or 10mg.
  For non-statin naive patients, regimens are to be changed to the equivalent dose of ezetimibe+rosuvastatin combination in case of already achieved LDL-cholesterol target (<70 mg/dL) and to be dosed up than the equivalent dose of study drugs in case of not yet achieved LDL-cholesterol target.
  Arms: Conventional-targeting group
Drug: Statin monotherapy (rosuvastatin or atorvastatin) — For statin naive patients, patients would initially receive Rosuvastatin 10 or 20mg or Atorvastatin 20 or 40mg. For non-statin native patients, regimens are to be change to equivalent dose of atorvastatin or rosuvastatin in case of already achieved LDL-cholesterol target (<70 mg/dL) and to be dosed up than the equivalent dose of study drugs in case of not yet achieved LDL-cholesterol target.
  Arms: Conventional-targeting group

SUMMARY:
Although the clinical efficacy of LDL-cholesterol lowering therapy has been proven with strong evidences and emphasized, there are also growing concerns that intensive lipid-lowering therapy would be related to increased risk of adverse effects. In addition, statin potency from recent guidelines was set from the studies composed of mainly Caucasian population, although there is an inconsistency of statin effect according to ethnicity. Asian population showed more profound LDL reduction not only from high potent statin but also from moderate to low potent statin. Conventional strategies for lowering LDL-cholesterol focused on statins, therefore doubling of previously described dose of statin would be common way in patients with inadequate LDL-cholesterol levels. Adding ezetimibe will be an alternative strategy not only to lower LDL-cholesterol level and also to reduce the need of dosage of high-intensity statin to achieve sufficient LDL-cholesterol lowering effect. However, studies regarding the effect of intensive-targeting of lipid-lowering therapy and therapy regimens are lacking. Thus, on these basis, we sought to evaluate whether intensive-targeting of lipid-lowering therapy will have more prominent beneficial effect compared to conventional-targeting in patients with documented ASCVD with either an ezetimibe/statin combination therapy or a statin monotherapy.

DETAILED DESCRIPTION:
All eligible patients who have documented ASCVD will be enrolled according to inclusion/exclusion criteria after voluntary agreement with informed consent. At the time of enrollment, we will stratify all patients according to LDL-cholesterol <100mg/dL, DM, and acute coronary syndrome, and randomly assign them in two groups according to LDL-cholesterol targeting level with a 1:1 ratio: "Intensive-targeting group" vs. "Conventional-targeting group". In addition, patients in each group will be randomly assigned to receive two lipid-lowering therapy regimen with a 1:1 ratio: "Ezetimibe/Statin combination therapy" vs. "Statin monotherapy". Patients allocated to each treatment group will receive lipid-lowering therapy with following protocols.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-80 years
2. Documented atherosclerotic cardiovascular disease (ASCVD)

   * Previous acute coronary syndrome (myocardial infarction [MI] or unstable angina),
   * Or stable angina with imaging or functional studies
   * Or coronary revascularization (percutaneous coronary intervention [PCI], coronary artery bypass graft [CABG], and other arterial revascularization procedures)
   * Or stroke and transient ischemic attack (TIA)
   * Or peripheral artery disease

Exclusion Criteria:

1. LDL-cholesterol level less than 70 mg/dL without statin therapyAllergy or hypersensitive to ezetimibe or statin
2. Active liver disease or persistent unexplained serum AST/ALT elevation more than 2 times the upper limit of normal range
3. Allergy or hypersensitivity to any statin or ezetimibe
4. Solid organ transplantation recipient
5. Pregnant women, women with potential childbearing, or lactating women
6. Life expectancy less than 3 years
7. Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
8. Inability to understand or read the informed content

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3048 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes by different lipid-lowering therapy | Within 3 years after the enrollment
  Composite of cardiovascular death, non-fatal MI, non-fatal stroke, any revascularization, and hospitalization for unstable angina

SECONDARY OUTCOMES:
Each component of primary endpoint within 3 years | Within 3 years after the enrollment
  * A. Rate of Cardiovascular death
  * B. Rate of non-fatal MI
  * C. Rate of non-fatal stroke
  * D. Rate of any revascularization
  * E. Rate of hospitalization for unstable angina
Various composite outcomes within 3 years | Within 3 years after the enrollment
  * A. Rate of composite of cardiovascular death, non-fatal MI, and non-fatal stroke
  * B. Rate of composite of cardiovascular death, non-fatal MI, non-fatal stroke, and any revascularization
  * C. Rate pf composite of cardiovascular death, non-fatal MI, and any revascularization
  * D. Rate of composite of all-cause death, non-fatal MI, non-fatal stroke, any revascularization, and hospitalization for unstable angina
Proportion of subjects achieving target LDL-cholesterol level | Within 3 years after the enrollment
Rate of cross-over into the non-allocated therapy regimen in order to achieve target LDL-cholesterol level | Within 3 years after the enrollment
Proportions of subjects requiring proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor to achieve target LDL-cholesterol level | Within 3 years after the enrollment
Difference in rate of primary outcome according to sex | Within 3 years after the enrollment
Difference in rate of primary outcome according to body mass index | Within 3 years after the enrollment
Rate of New-onset diabetes mellitus | Within 3 years after the enrollment
Rate of worsening of glycemic control or homeostatic model assessment (HOMA)-index | Within 3 years after the enrollment
Occurrence of statin-associated muscle symptoms (SAMS) requiring change of therapy regimen or dosage | Within 3 years after the enrollment
Occurence of elevation of muscle enzymes (CPK > 4 x UNL) | Within 3 years after the enrollment
Occurence of elevation of hepatic enzymes (AST, ALT, or both ≥ 3 x UNL) | Within 3 years after the enrollment
Occurence of elevation of serum creatinine level (>50% from baseline) | Within 3 years after the enrollment
Change of proteinuria | Within 3 years after the enrollment
Rate of cancer diagnosis | Within 3 years after the enrollment
Rate of operation due to cataract | Within 3 years after the enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No